CLINICAL TRIAL: NCT04600076
Title: MOMSonLINE2:A Pilot Study Testing Recruitment and Retention of Women of Color to an Online Support Group for Bereaved Mothers
Brief Title: MOMSonLINE2 ; A Pilot Study Testing Recruitment and Retention of Women of Color to an Online Support Group for Bereaved Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Katherine Gold, Associate Professor of Family Medicine and Associate Professor of Obstetrics and Gynecology, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00159800; UL1TR002240 (NIH)
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Results first posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Stillbirth; Grief; Infant Death
Keywords: internet support site; BabyCenter.com.
MeSH Terms: conditions — Stillbirth; Infant Death

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BabyCenter site and the community group (Experimental)
  Interventions: Behavioral: BabyCenter site and the community group

INTERVENTIONS:
Behavioral: BabyCenter site and the community group — Participants will be asked to sign on to the BabyCenter community group for people with pregnancy or infant loss at least 3 times weekly for 6 weeks. Participants may choose to post or comment on the site but are not required to do so.

SUMMARY:
This is a 6-week pilot study to see how research participants feel about an internet support site after a stillbirth or infant death. Losing a baby through stillbirth or early infant death is typically devastating for families. However, investigators do not know if internet on-line support for parents helps manage grief more easily.

In addition to using the BabyCenter.com website, participants will be asked to complete online surveys at the beginning and the end of the study, as well partake in an interview.

Data from this pilot study will help develop a much larger randomized control study of on-line support outcomes after perinatal loss.

ELIGIBILITY:
Inclusion Criteria:

* Michigan residence and infant delivery
* Non-Caucasian race and/or Hispanic ethnicity
* Read/speak English
* Gave birth to a stillborn baby or had an infant death in the first 28 days of life
* Did not give the baby up for adoption pre-loss
* Internet access

Exclusion Criteria:

* Don't Read/speak English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gave birth to a stillborn baby or had an infant death in the first 28 days of life. Age 18 or older at delivery.
Enrollment: 22 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Gold, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gold KJ, Dobson ML, Sen A. "Three Good Things" Digital Intervention Among Health Care Workers: A Randomized Controlled Trial. Ann Fam Med. 2023 May-Jun;21(3):220-226. doi: 10.1370/afm.2963. PMID 37217328
- [Derived] Gold KJ, Boggs ME, Plegue MA, Andalibi N. Online Support Groups for Perinatal Loss: A Pilot Feasibility Study for Women of Color. Cyberpsychol Behav Soc Netw. 2022 Aug;25(8):534-539. doi: 10.1089/cyber.2021.0304. Epub 2022 Jul 20. PMID 35861706

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BabyCenter Site and the Community Group
Started | 22
Completed | 19
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | BabyCenter Site and the Community Group
Number analyzed (Participants) | 22
Age, Continuous [Mean (Full Range); unit: years] | 31 [21 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 3
  More than one race | 4
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Approached for Enrollment Who Signed up for the Study
Description: Feasibility of recruitment as shown by percent of those approached for enrollment who signed up for the study.
Time Frame: 6 months
Population: This is the total number of potential participants who were actually invited to be included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | BabyCenter Site and the Community Group
Number analyzed (Participants) | 200
Participants | 22

2. Primary Outcome: Feasibility: Retention
Description: Number of participants that completed:
  * The 6 week intervention.
  * Pre-post surveys.
  * Phone interview
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | BabyCenter Site and the Community Group
Number analyzed (Participants) | 22
Participants
  6 week intervention | 20
  Pre-post surveys | 20
  Phone interview | 19

3. Secondary Outcome: Change in Depression as Measured by The Personal Health Questionnaire Depression (PHQ-8)
Description: The Personal Health Questionnaire Depression (PHQ-8) is a widely used and validated screen for depression. The PHQ-8 is scored by adding scores from each question (0-3) to a final score (0 to 24). Higher scores indicate worse outcome and a score of 10 or higher indicates a positive screen. A positive screen is probable for clinical depression.
Time Frame: Pre intervention (day 0), Post intervention (6 weeks)
Population: Only 17 participants answered all pre and post intervention survey depression questions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BabyCenter Site and the Community Group
Number analyzed (Participants) | 17
score on a scale
  Pre-Intervention PHQ-8 | 9.1 (6.4)
  Post-Intervention PHQ-8 | 8.1 (5.2)

4. Secondary Outcome: Change in Post-traumatic Stress Disorder (PTSD)
Description: PTSD will be measured using the 20-question Post-traumatic stress disorder (PTSD) checklist for the Diagnostic and Statistical Manual of Mental Disorders (DSM) -5 (PTSD Checklist for DSM-5, Civilian Version). Scores range from 0-80. A score of 33 or above will be used as our cutoff. A score above this indicated a probable diagnosis of PTSD.
Time Frame: Pre intervention (day 0), Post intervention (6 weeks)
Population: Of all the participants who completed, analysis covers only those who answered all questions on pre and post surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BabyCenter Site and the Community Group
Number analyzed (Participants) | 18
score on a scale
  Pre-Intervention PTSD | 38.6 (14.9)
  Post-Intervention PTSD | 35.8 (13.6)

5. Secondary Outcome: Change in Anxiety Based on the Generalized Anxiety Disorder Screen (GAD-7)
Description: The Generalized Anxiety Disorder screen (GAD-7) is a seven-item self-report instrument for screening, diagnosis and severity assessment of anxiety disorder. The GAD-7 total score for the seven items ranges from 0 to 21: 0-4 Minimal anxiety; 5-9 Mild anxiety; 10-14 Moderate anxiety; 15-21 Severe anxiety.
Time Frame: Pre intervention (day 0), Post intervention (6 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BabyCenter Site and the Community Group
Number analyzed (Participants) | 19
score on a scale
  Pre-Intervention GAD-7 | 12.8 (5.7)
  Post-Intervention GAD-7 | 11.9 (5.6)

6. Secondary Outcome: Change in Grief Based on the Perinatal Grief Scale
Description: The Perinatal Grief Scale measures grief, coping, and despair following the death of a child. It includes 33 questions on a 5-point Likert scale that ranges from 1=strongly agree to 5=strongly disagree. A higher score would indicate more grief and a lower score less grief. A score cutoff of >40 to indicates more severe grief. Two questions were inadvertently dropped from the PGS in our surveys; this allows pre-post analysis but limits comparison to other studies. With this omission, our PGS scores could range from 31 -155.
Time Frame: Pre intervention (day 0), Post intervention (6 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BabyCenter Site and the Community Group
Number analyzed (Participants) | 19
score on a scale
  Pre-Intervention PGS | 91.9 (18.9)
  Post-Intervention PGS | 88.1 (19.7)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | BabyCenter Site and the Community Group
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-18): https://cdn.clinicaltrials.gov/large-docs/76/NCT04600076/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-24): https://cdn.clinicaltrials.gov/large-docs/76/NCT04600076/ICF_001.pdf